CLINICAL TRIAL: NCT01496248
Title: The Effect of Korean Red Ginseng as Adjuvant Treatment for the Residual Symptoms of Depression
Brief Title: Efficacy Study of Korean Red Ginseng to Treat Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Young-Hoon Ko, Associate Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1105721
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Residual symptoms; Korean red ginseng
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Korean Red Ginseng (Experimental): Extract of Korean red ginseng was administrated to subjects through capsule form.
  Interventions: Dietary Supplement: Korean Red Ginseng

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — 100% of the past psychiatric medication dose will be maintained during 8 week study period. Korean Red ginseng will be started with 2g/day and then maintained using flexible dosing of 2-3g/day during the study period.

SUMMARY:
The purpose of this study is to determine whether Korean Red Ginseng are effective in the treatment of the residual symptoms of depression as an adjuvant treatment.

DETAILED DESCRIPTION:
Thirty-five female outpatients aging from 18 to 65 years, who were remitted from major depression with residual symptoms (Montgomery Asberg Depression Rating Scale, MADRS ≤ 12), were given Korean red ginseng at doses of 3g / day during 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who met Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for major depressive disorder.
* Those who are in remission, which is defined as a MADRS score 8 on two consecutive visits at a 4-week interval.
* Their primary psychiatric clinician determined that they would benefit from an adjuvant treatment of Korean red ginseng for residual symptoms.

Exclusion Criteria:

* Those who have a history of substance abuse or dependence within 1 month.
* Those who have clinically significant abnormal laboratory values or any other abnormal baseline laboratory findings considered by psychiatrists to be indicative of conditions that might affect the study results.
* Those who have a past history of hypersensitivity or intolerance to Korean red ginseng.
* Those who participated in clinical trials within 1 month before entering the study entry.
* Those who are pregnant or are breast feeding.
* Those who have a immediate risk of harming self or others or history of suicide attempts in the year before the screening precluded inclusion in the study.
* The patients unable/unlikely to comprehend/follow the protocol.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Ko, M.D., Ph.D., Principal Investigator — Korea University Medical Centre
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Jeong HG, Ko YH, Oh SY, Han C, Kim T, Joe SH. Effect of Korean Red Ginseng as an adjuvant treatment for women with residual symptoms of major depression. Asia Pac Psychiatry. 2015 Sep;7(3):330-6. doi: 10.1111/appy.12169. Epub 2014 Dec 12. PMID 25504813

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Korean Red Ginseng
Started | 35
Completed | 25
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 35

OUTCOME MEASURES:

1. Primary Outcome: Depression Residual Symptom Scale
Description: This consists of 25 items and includes specific residual depressive symptoms, e.g. sadness and anhedonia, lack of energy, psychomotor retardation and anxiety, as well as items reflecting subjective feelings of vulnerability, loss of internal reference points and increased emotionalism. Patients were instructed to compare the past 7 days with the period before the very first symptoms of the most recent depressive episode. Each item is scored as 0 to 3. A total score is the range from 0(none) to 75(most severe).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 21.8 (12.7)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Depression Residual Symptom Scale
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 17.5 (11.1)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Visual Analogue Scale
Description: This has been described as simple, highly sensitive, and reliable rating scales for subjective experiences. The VAS in this study is used for assessing of variation in severity of residual symptoms. The subject is asked to indicate his/her perceived symptom severity along a 100 mm horizontal line, and this rating is then measure from the left edge (0, no symptom) to right edge (100, most severe).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 31.4 (22.1)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: Visual Analogue Scale
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 28.0 (26.5)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

5. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: This is a 10-item depression rating scale, widely used in depressed patients. Each item is rated from 0 to 6. A total score is the range from 0(none) to 60(most severe). The MADRS has been designed to measure severity of depression in clinical samples and be sensitive to change during antidepressant treatment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 6.7 (2.7)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

6. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: as for outcome 5
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 4.4 (3.1)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: Clinical Global Index
Description: This was developed for use in psychopharmacology trials and then, it has been expanded in its use as a standard primary measure in studies investigating the efficacy of pharmacological treatments for various psychiatric illnesses such as depression, anxiety disorder, and bipolar disorder. The CGI-S rates the severity of the patient's illness, on a 7-point scale ranging from 1(Normal) 1 to 7(Extremely ill), according to the clinician's experience of patients suffering from the same condition.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 3.1 (0.5)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Clinical Global Index
Description: as for outcome 7
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Korean Red Ginseng
Number analyzed (Participants) | 25
units on a scale | 2.4 (0.5)
Statistical Analysis 1: Comparison: Korean Red Ginseng; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Korean Red Ginseng
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 5/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Korean Red Ginseng (N=35)
headache (Nervous system disorders) | 4 (4)
sleep problem (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No